CLINICAL TRIAL: NCT04675021
Title: A Phase I Open-label Study to Assess the Absolute Bioavailability of Savolitinib and Absorption, Distribution, Metabolism, Excretion of [14C]Savolitinib in Healthy Male Subjects
Brief Title: Absolute Bioavailability and ADME Study of Savolitinib in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Quotient Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D5084C00010
Record Dates: First submitted 2020-11-12; First posted 2020-12-19 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Cancer
Keywords: Cancer
MeSH Terms: conditions — Neoplasms | interventions — 1-(1-(imidazo(1,2-a)pyridin-6-yl)ethyl)-6-(1-methyl-1H-pyrazol-4-yl)-1H-(1,2,3)triazolo(4,5-b)pyrazine; Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AZD6094 (Savolitinib) D5084C00010 (Experimental): All volunteers will receive either a single dose or two doses of AZD6094 (Savolitinib) D5084C00010
  Interventions: Drug: AZD6094 (Savolitinib) film coated tablets 600 mg; Drug: [14C]-AZD6094 (Savolitinib) Solution for Infusion, 20 μg/mL (NMT 37.0 kBq/5 mL); Drug: [14C] AZD6094 (Savolitinib) Oral Solution, 300 mg (NMT 4.1 MBq)

INTERVENTIONS:
Drug: AZD6094 (Savolitinib) film coated tablets 600 mg — AZD6094 (Savolitinib) ilm Coated Tablet 200 mg x 3
  Other Names: AZD6094 (Savolitinib) Film Coated Tablet 200 mg x 3
Drug: [14C]-AZD6094 (Savolitinib) Solution for Infusion, 20 μg/mL (NMT 37.0 kBq/5 mL) — 14C AZD6094 (Savolitinib) Solution for Infusion (20 μg/mL (NMT 37.0 kBq/5 mL)
  Other Names: 14C AZD6094 (Savolitinib) Solution for Infusion (20 μg/mL (NMT 37.0 kBq/5 mL)
Drug: [14C] AZD6094 (Savolitinib) Oral Solution, 300 mg (NMT 4.1 MBq) — 14CAZD6094 (Savolitinib) Oral Solution (300 mg NMT 4.1MBq)
  Other Names: 14CAZD6094 (Savolitinib) Oral Solution (300 mg NMT 4.1MBq)

SUMMARY:
The Sponsor is developing the test medicine, AZD6094 (Savolitinib) for the potential treatment of cancer. Cancer is a condition where cells in a specific part of the body grow and reproduce uncontrollably, causing a growth called a tumour. The test medicine works to inhibit a pathway within the body which promotes tumours to grow and spread. The study involves radiolabelling (labelling the molecule with radioactive 14C) which is used to locate the molecule within the body.

The study will evaluate the absolute bioavailability of the test medicine (amount of the oral test medicine that enters the blood stream relative to the dose given into the vein), along with the mass balance (how much radioactivity can be recovered from the urine and faeces) and the rates and routes of elimination of [14C]savolitinib. It will also look to identify the breakdown products (metabolites) of the test medicine. The safety and tolerability of the test medicine will be assessed.

The study will consist of two parts, involving a minimum of eight healthy male volunteers. In Part one, following a high fat breakfast, volunteers will receive a single oral dose of the test medicine, followed by an intravenous infusion (solution into the vein) of radiolabelled test medicine. Volunteers will remain resident in the clinical unit until 72 hours post-oral dose.

There will then be a washout period of at least 14 days, after which the volunteers will return to the clinical unit for Part two. Volunteers will receive a single oral dose of radiolabelled test medicine as an oral solution. Blood, urine and faecal samples will be collected from volunteers whilst they are resident in the clinical unit for up to 168 hours postdose (Day 8). Volunteers will return for a follow-up visit at least 14 days after their last dose for safety assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study specific procedures.
2. Healthy male subjects aged 30 to 65 years at the time of signing informed consent with suitable veins for cannulation or repeated venepuncture.
3. Body mass index (BMI) of 18.0 to 32.0 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive, as measured at screening.
4. Must be willing and able to communicate and participate in the whole study
5. Must have regular bowel movements (i.e., average stool production of ≥1 and

   ≤3 stools per day).
6. Adequate coagulation parameters, defined as: International Normalisation Ratio (INR) <1.5 x ULN and activated partial thromboplastin time (aPTT) <1.5 x ULN.
7. Must agree to adhere to the contraception requirements defined in Section 9.4. Subjects aged under 45 years must have had a vasectomy. Subjects must be willing to agree to not father children for a further 6 months after the study follow-up visit.

Exclusion Criteria:

1. History of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate in the study.
2. History or presence of GI, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
3. Acute diarrhoea or constipation in the 7 days before administration of IMP in the study. If screening occurs >7 days before the first study day, this criterion will be determined on first study day.
4. Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of IMP.
5. Any clinically significant abnormalities in clinical chemistry, haematology, or urinalysis results, as judged by the investigator. Subjects with Gilbert's Syndrome are not allowed.
6. Any clinically significant abnormal findings in vital signs, as judged by the investigator.
7. Any clinically significant abnormalities on 12-lead ECG, as judged by the investigator. Mean resting corrected QT interval (QTcF) >450 msec on screening or pre-dose (Part 1 only) obtained from 3 ECGs or factors that may increase the risk of QTcF prolongation or any clinically important abnormalities in rhythm, conduction or morphology of resting electrocardiograms (ECGs), e.g., complete left bundle branch block, third degree heart block, second degree heart block, PR interval >250 msec.
8. Any factors that may increase the risk of QTcF prolongation such as chronic hypokalaemia not correctable with supplements, congenital or familial long QT syndrome, or family history of unexplained sudden death under 40 years of age in first-degree relatives or any concomitant medication known to prolong the QT interval and cause Torsade de Pointes.
9. Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody, and human immunodeficiency virus (HIV) antibody.
10. Known or suspected history of drug abuse, as judged by the investigator.
11. Has received another new chemical entity (defined as a compound which has not been approved for marketing; including radiolabelled chemical entity) within 90 days or five elimination half-lives, whichever is longer, of the first dosing date in this study. The period of exclusion lasts for 90 days or five elimination halflives after the final dose or 1 month after the last visit, whichever is the longest. Note: subjects consented and screened, but not administered IMP in this study or a previous Phase I study, are not excluded
12. Plasma donation within 1 month of screening or any blood donation/loss more than 500 mL during the 3 months prior to screening.
13. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the investigator or history of hypersensitivity to drugs with a similar chemical structure or class to savolitinib. Hay fever is allowed unless it is active
14. Evidence of current SARS-CoV-2 infection.
15. History of any alcohol abuse in the past 2 years.
16. Regular alcohol consumption in males >21 units per week (1 unit = ½ pint beer, or a 25 mL shot of 40% spirit, 1.5 to 2 Units = 125 mL glass of wine, depending on type).
17. Current smokers or those who have smoked or used nicotine products (including e-cigarettes) within the 6 months prior to screening. A confirmed breath carbon monoxide reading of greater than 10 ppm at screening or admission.
18. Subjects with pregnant or lactating partners.
19. Radiation exposure, including that from the present study, excluding background radiation but including diagnostic x-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 2017 [9], shall participate in the study.
20. Subjects who have been administered IMP in an 14C ADME study in the last 12 months.
21. Subjects with a history of cholecystectomy or gall stones.
22. Positive screen for drugs of abuse or alcohol at screening or on each admission to the study centre.
23. Subjects with estimated glomerular filtration rate [eGFR] of <60 mL/min/1.73m2, as measured at screening, using the chronic kidney disease epidemiology collaboration (CKD-EPI) equation, or evidence of renal impairment in subjects with eGFR between 60 and 90 mL/min/1.73m2.
24. Subjects with a presence of any of the following at screening:

    <LLN for haemoglobin value, WBC, neutrophil count, lymphocytes and platelet count
25. Total bilirubin, ALT/AST>ULN at screening.
26. Use of drugs with enzyme-inducing properties such as St John's Wort within 3 weeks prior to the first administration of IMP.
27. Use of any prescribed or nonprescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the two weeks prior to the first administration of IMP or longer if the medication has a long half-life.
28. Excessive intake of caffeine-containing drinks or food (e.g., coffee, tea, chocolate) as judged by the investigator. Excessive intake of caffeine defined as the regular consumption of more than 600 mg of caffeine per day (e.g., >5 cups of coffee) or would likely be unable to refrain from the use of caffeine-containing beverages during confinement at the investigational site.
29. Involvement of any AstraZeneca, Quotient or study site employee or their close relatives.
30. Subjects who report to have previously received savolitinib.
31. Judgment by the investigator that the volunteer should not participate in the study if they have any ongoing or recent (i.e., during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements.
32. Subjects who cannot communicate reliably with the investigator.
33. Vulnerable subjects, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.
34. Non-leukocyte depleted whole blood transfusion within 120 days of the date of the genetic sample collection or previous bone marrow transplant.
35. History of latent or chronic infections (e.g., tuberculosis, recurrent sinusitis, genital herpes, recurrent urinary tract infections) or at risk of infection (surgery, trauma or significant infection within previous 90 days, history of skin abscesses within previous 90 days prior to first IMP dose).
36. Planned in-patient surgery, dental procedure or hospitalisation during the study.
37. Failure to satisfy the investigator of fitness to participate for any other reason.

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Healthy male subjects aged 30 to 65 years at the time of signing informed consent
Enrollment: 8 (Actual)
Dates: Start 2020-11-13 (Actual); Primary Completion 2021-01-11 (Actual); Study Completion 2021-01-11 (Actual)

PRIMARY OUTCOMES:
Absolute Bioavailability (F) of savolitinib | Collection of plasma samples from pre-dose to 72 hours post-dose
  Absolute bioavailability based on AUC0-inf of oral formulation compared to IV adjusted for dose
The cumulative amount of AZD6094 (savolitinib) excreted (CumAe) | Urine and faecal samples collected from pre-dose until 168 hours post-dose
  Assessment of the total radioactivity by measuring the cumulative amount of AZD6094 (savolitinib) excreted (CumAe)
The cumulative amount of AZD6094 (savolitinib) excreted and expressed as a percentage of the administered dose (CumFe) | Urine and faecal samples collected from pre-dose until 168 hours post-dose
  Assessment of the total radioactivity by measuring the cumulative amount of AZD6094 (savolitinib) excreted and expressed as a percentage of the administered dose (CumFe)
Assessment of metabolites in plasma by liquid chromatography-radiochemical-detection and subsequent mass spectrometry | Plasma samples collected until 168 hours post-dose
  Assessment of metabolites in plasma by liquid chromatography-radiochemical-detection and subsequent mass spectrometry
Assessment of metabolites in urine by liquid chromatography-radiochemical-detection and subsequent mass spectrometry | Urine samples collected until 168 hours post-dose
  Assessment of metabolites in urine by liquid chromatography-radiochemical-detection and subsequent mass spectrometry
Assessment of metabolites in faeces by liquid chromatography-radiochemical-detection and subsequent mass spectrometry | Faeces samples collected until 168 hours post-dose
  Assessment of metabolites in faeces by liquid chromatography-radiochemical-detection and subsequent mass spectrometry

SECONDARY OUTCOMES:
Number of AE's experienced by subjects | AEs recorded from the time of informed consent until the follow up visit (approx 10 weeks)
  Safety and tolerability assessed through the incidence of AEs
Time to maximum concentration (tmax) for AZD6094 (savolitinib) and total radioactivity | Collection of plasma samples from pre-dose to 168 hours post-dose
  Assessment of pharmacokinetics of AZD6094 (savolitinib) and total radioactivity by measuring the time to maximum concentration (tmax)
Maximum observed concentration for AZD6094 and total radioactivity | Collection of plasma samples from pre-dose to 168 hours post-dose
  Assessment of pharmacokinetics of AZD6094 and total radioactivity by measuring the maximum observed concentration (cmax)
Area under the curve from time 0 to the time of last measurable concentration for AZD6094 (savolitinib) and total radioactivity | Collection of plasma samples from pre-dose to 168 hours post-dose
  Assessment of pharmacokinetics of AZD6094 (savolitinib) and total radioactivity by measuring the area under the curve from time 0 to the time of last measurable concentration
Area under the curve from time 0 extrapolated to infinity for AZD6094 (savolitinib) and total radtioactivity | Collection of plasma samples from pre-dose to 168 hours post-dose
  Assessment of pharmacokinetics of AZD6094 (savolitinib) and total radioactivity by measuring the area under the curve from time 0 extrapolated to infinity
Terminal elimination half-life for AZD6094 (savolitinib) and total radioactivity | Collection of plasma samples from pre-dose to 168 hours post-dose
  Assessment of pharmacokinetics of AZD6094 (savolitinib) and total radioactivity by measuring the terminal elimination half-life
First order rate constant associated with the terminal (log-linear) portion of the curve for AZD6094 (savolitinib) and total radioactivity | Collection of plasma samples from pre-dose to 168 hours post-dose
  Assessment of pharmacokinetics of AZD6049 (savolitinib) and total radioactivity by measuring the First order rate constant associated with the terminal (log-linear) portion of the curve
Total body clearance calculated after a single extravascular administration for AZD6094 (savolitinib) and total radioactivity | Collection of plasma samples from pre-dose to 168 hours post-dose
  Assessment of pharmacokinetics of AZD6049 (savolitinib) and total radioactivity by measuring the total body clearance calculated after a single extravascular administration
Apparent volume of distribution based on the terminal phase for AZD6094 (savolitinib) and total radioactivity | Collection of plasma samples from pre-dose to 168 hours post-dose
  Assessment of pharmacokinetics of AZD6049 (savolitinib) and total radioactivity by measuring the apparent volume of distribution based on the terminal phase
Renal clearance for AZD6094 (savolitinib) and total radioactivity | Collection of plasma samples from pre-dose to 168 hours post-dose
  Assessment of pharmacokinetics of AZD6049 (savolitinib) and total radioactivity by measuring the renal clearance
Evaluation of whole blood to plasma concentration ratios for total radioactivity | Collection of blood samples until 168 hours post dose
  Assessment of total radioactivity in whole blood and plasma

OTHER OUTCOMES:
Identification of the chemical structure of major metabolite(s) in plasma | Plasma samples collected until 168 hours post-dose
  Quantification and identification of the chemical structures of metabolites of AZD6094 (savolitinib)
Identification of the chemical structure of major metabolite(s) in urine | Urine samples collected until 168 hours post-dose
  Quantification and identification of the chemical structures of metabolites of AZD6094 (savolitinib)
Identification of the chemical structure of major metabolite(s) in faeces | Faeces samples collected until 168 hours post-dose
  Quantification and identification of the chemical structures of metabolites of AZD6094 (savolitinib)
Collection and storage of DNA for future exploratory research | A maximum of 15 years following the last subject's last visit in the study
  Collect and store DNA for future exploratory research into genes/genetic variations that may influence the PK of savolitinib

CONTACTS AND LOCATIONS:
Overall Officials: Somasekhara Menakuru, MBBS MS MRCS, Principal Investigator — Quotient Sciences
Locations (1):
- Research Site, Ruddington, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the AZ approved data access tool to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Miah K, Vishwanathan K, Scarfe G, Li Y, Hara I, Cantarini M, Argue J, Menakuru SR. A Phase 1 Study to Evaluate Absolute Bioavailability and Absorption, Distribution, Metabolism, and Excretion of Savolitinib in Healthy Male Volunteers. Clin Pharmacol Drug Dev. 2023 Apr;12(4):424-435. doi: 10.1002/cpdd.1224. Epub 2023 Feb 19. PMID 36808891